CLINICAL TRIAL: NCT06276634
Title: Intermittent Hypoxia Initiated Motor Plasticity in Individuals With Multiple Sclerosis
Brief Title: Intermittent Hypoxia in Persons With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Northwestern University (Other)
Responsible Party: Principal Investigator, Milap Sandhu, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU00219535; R21HD108587 (NIH)
Record Dates: First submitted 2023-12-11; First posted 2024-02-26 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis-Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive
Keywords: multiple sclerosis; AIH; Hypoxia
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Hypoxia | interventions — Insemination, Artificial, Homologous

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, cross-over, repeated measures study design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AIH First (Experimental): Participants in the AIH First arm will undergo 5 days of Acute Intermittent Hypoxia Interventions. Following the 5 Days of AIH, after a 2-week washout period, this group will then undergo 5 days of Sham AIH Interventions. The procedures are identical to AIH but with 21% oxygen for both breath cycles
  Interventions: Other: Acute Intermittent Hypoxia; Other: Sham-Acute Intermittent Hypoxia
- Sham First (Experimental): Participants in the Sham First arm will undergo 5 days of Sham-Acute Intermittent Hypoxia Interventions. Following the 5 Days of Sham-AIH, after a 2-week washout period, this group will then undergo 5 days of AIH Interventions. The procedures are identical to Sham-AIH but with 9-10% oxygen for the first breath cycle
  Interventions: Other: Acute Intermittent Hypoxia; Other: Sham-Acute Intermittent Hypoxia

INTERVENTIONS:
Other: Acute Intermittent Hypoxia — During each AIH session, the participant will be equipped with a non-rebreathing face mask, and provided with the AIH intervention. The AIH intervention involves alternating breathing cycles: one with lower oxygen concentration (9-10% Oxygen) than that at sea level (~21% Oxygen) lasting between 30 and 60 seconds, followed by a similar duration of normal room air (21% Oxygen). This cycle will be repeated 15 times in one session, continuous blood oxygen levels and heart rate will be monitored.
  Other Names: AIH
Other: Sham-Acute Intermittent Hypoxia — During each Sham-AIH session, the participant will be equipped with a non-rebreathing face mask, and provided with the Sham-AIH intervention. The Sham-AIH intervention involves alternating breathing cycles: both with oxygen concentrations of ~21% Oxygen lasting between 30 and 60 seconds, followed by another similar duration of normal room air (21% Oxygen). This cycle will be repeated 15 times in one session, continuous blood oxygen levels and heart rate will be monitored.

SUMMARY:
This study aims to understand the mechanisms of a novel intervention involving breathing short durations of low levels of oxygen for persons with multiple sclerosis (MS). This intervention with low levels of oxygen is called Acute Intermittent Hypoxia (AIH), the levels of oxygen experienced are similar to breathing the air on a tall mountain, for less than 1 minute at a time. Previous studies have shown that AIH is a safe and effective way to increase strength in persons with MS. Here the investigators aim to look at brain activation and ankle strength before and after AIH to gain a better understanding of how the AIH may improve strength in those persons with MS.

DETAILED DESCRIPTION:
Recent research has shown that AIH, characterized by brief episodes of reduced oxygen levels in the inspired air, has the potential to induce neural adaptations. These adaptations are suspected to influence several aspects of neuroplasticity, including the modulation of neurotransmitters and neurotrophic factors. Persons with MS typically exhibit greater cortical activation to achieve a given motor task compared to healthy controls, suggesting compensatory activations in motor cortices and the recruitment of additional non-motor regions for successful motor control. Therefore, interventions that promote adaptive neuroplasticity in motor control systems may induce a reduction in fMRI activation during motor tasks as well as an increase in functional connectivity between somatomotor cortices. This study will explore potential mechanisms of this intervention in MS using motor task performance and advanced neuroimaging techniques.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of relapsing form of MS (including relapsing-remitting MS and secondary-progressive MS)
* Expanded Disability Status Scale (EDSS) score of at least 3 and no more than 6.5
* Motor Functional System Scale (FSS) between 2-4
* Relapse free for at least 1 year
* Age ≥ 18 years and ≤ 75 years
* Safe to be scanned based on MRI questionnaire
* Participants using dalfampridine will be eligible if taking the same daily dose for at least 2 months prior to screening

Exclusion Criteria:

* Active contrast-enhancing MS lesions, or diffusion positive lesions suggestive of acute cerebrovascular disease on baseline MRI scan
* Uncontrolled hypertension (Systolic between 85 and 140, diastolic between 90 and 55)
* History of epilepsy
* Chronic obstructive pulmonary disease
* Uncontrolled Sleep apnea
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Ankle Plantarflexion Strength | Before and following each 5-day intervention block
  Participants will be seated in an adjustable chair with tested foot secured to a foot plate with the ankle in line with a rotational load cell. Participants will be asked to produce maximal ankle plantarflexion contractions, Electromyographic signals of the gastrocnemius, tibialis anterior, and soleus will be recorded simultaneously

SECONDARY OUTCOMES:
Task fMRI | Before and following each 5-day intervention block
  This outcome observes neural activations during voluntary muscle activations

OTHER OUTCOMES:
Timed 25 Feet Walk test | Before and following each 5-day intervention block
  A part of the MS functional composite. Participants will be directed to walk across a 25-foot course as quickly and safely as possible.
Six-Minute Walk test | Before and following each 5-day intervention block
  The Six-minute walk test is an assessment to measure the distance able to be traversed by a participant in 6-minutes
Stride length | Before and following each 5-day intervention block
  This assessment involves walking at normal walking pace over flat ground. The GAITRite®, a pressure sensitive walkway, will be used to measure and analyze spatiotemporal gait parameters, particularly stride length in meters
12-Item Multiple Sclerosis walk scale (MSWS-12) | Before and following each 5-day intervention block
  This is a self-reported measure of the impact of MS on an individual's walking ability Minimum score: 12 Maximum score: 60 A lower score indicates better walking ability, less affected by the multiple sclerosis
Resting-State fMRI | Before and following each 5-day intervention block
  Participants will undergo an 2D T2* weighted multi-band multi-echo gradient echo-planar imaging sequence at rest

CONTACTS AND LOCATIONS:
Overall Officials: Milap Sandhu, Pt, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
We do not currently have a plan to share IPD